CLINICAL TRIAL: NCT06636318
Title: Impact of a 24-hour Shift Call on the Immune Status of Surgery Residents
Brief Title: Immune Status After Being on Call for 24 Hrs
Status: Recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: IRB24-1426
Record Dates: First submitted 2024-09-27; First posted 2024-10-10 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Sleep Deprivation
MeSH Terms: conditions — Sleep Deprivation | interventions — Monitoring, Physiologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- General Surgery Residents: General Surgery residents on during 24-hour rotation shifts
  Interventions: Diagnostic Test: Blood Sample Collection; Device: Actigraph (GT9X-BT) Monitor

INTERVENTIONS:
Diagnostic Test: Blood Sample Collection — To characterize the phenotype and function of immune cells in surgery residents before and after a 24-hour shift, and before and after a month of being "on call". Along with to investigate the relationship between sleep deprivation, physical activity, and different immune responses.
Device: Actigraph (GT9X-BT) Monitor — Participants will be asked to wear their monitor every day for a week. The monitor will collect their step count, sleep and heart rate automatically. Participants will return their monitor at visit 5 (day 30) of the study.

SUMMARY:
Sleep deprivation is a prevalent problem in modern societies. Sleep deprivation can cause hormonal changes, such as an increase in cortisol, as well as inflammation. Animal studies have shown an increase in inflammatory cytokine production following sleep deprivation. Additionally, humans experiencing sleep deprivation may experience a decrease in natural killer cells and lymphocytes.

Physicians, particularly those in surgical specialties, are often subjected to sleep deprivation as part of their medical residency training. This study hypothesizes that after 24-hour shifts, there is an increase in inflammatory response and impairment of the immune response against unspecific activation. This proposal aims to provide insight into the impact of sleep deprivation on the immune system of surgery residents by characterizing the phenotype and function of immune cells, as well as their correlation with biometric data.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Surgery residents in a 24-hour shift rotation
* Gender of subjects: Males and females
* Age of subjects: 18 years old and older
* Racial and Ethnic Origin: Any race or ethnicity

Exclusion Criteria:

* Unwilling/unable to sign informed consent
* Vulnerable Subjects/Subject Capacity to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General Surgery residents, on during 24-hour shifts
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Characterization of the phenotype and function of immune cells using flow cytometry | 24 hours
  Specifically, T cells, B cells, dendritic cells, macrophages, and natural killer cells will be identified and analyzed. Memory cells, co-inhibitor markers, and regulatory markers will also be evaluated. The function will be analyzed based on the intracellular expression of effector molecules and cytokines after unspecific activation with CD3-CD28 beads.

SECONDARY OUTCOMES:
Analyze the biometric data and correlate it with changes in sleep deprivation | One week before rotation and the last week of rotation
  To examine the associations, participants will be using an activity and sleep monitor.
Analyze the biometric data and correlate it with changes in the immune response | One week before rotation and the last week of rotation
  To examine the associations, participants will be using an activity and sleep monitor.
Analyze the biometric data and correlate it with changes in physical activity | One week before rotation and the last week of rotation
  To examine the associations, participants will be using an activity and sleep monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Angelica Perez-Gutierrez, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No